CLINICAL TRIAL: NCT03962920
Title: Personalized Treatment of Urogenital Cancers Depends on the Microbiome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZUHURO
Record Dates: First submitted 2019-05-23; First posted 2019-05-24 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Microbial Disease
MeSH Terms: interventions — Tigecycline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical treatment + antibiotics (Active Comparator): Use antibiotic
  Interventions: Drug: Tigecycline 50 MG
- surgical treatment + placebo (Placebo Comparator): Use placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tigecycline 50 MG — Local instillation of drug directly to the tumour tissue
  Other Names: Tigecycline
  Arms: Surgical treatment + antibiotics
Other: Placebo — Local instillation of sterile water directly to the tumour tissue
  Other Names: Sterile water
  Arms: surgical treatment + placebo

SUMMARY:
This is a randomized controlled trial where patients undergoing surgical treatment for urogenital cancers will be randomized in a two arms study: surgical treatment + antibiotics OR surgical treatment + placebo.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy verified diagnosis of urological cancer, localized disease

Exclusion Criteria:

* Hospitalization within three months of surgery
* Antibiotics within three months of surgery
* Infectious disease, including UTI's within three months of surgery
* History of cancers of the genitourinary tract
* Diabetes

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
recurrence rate after surgical treatment of tumour | 5 years after treatment
  recurrence rate after surgical treatment of tumour

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University Hospital, Roskilde, Denmark